CLINICAL TRIAL: NCT03324256
Title: Acute Effect of Energy Drinks on Vascular Function
Brief Title: Energy Drinks and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB201700678
Record Dates: First submitted 2017-10-20; First posted 2017-10-27 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Vascular Function
Keywords: Energy drink consumption
MeSH Terms: interventions — Energy Drinks

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Energy drink and placebo gum (Active Comparator): Commercially-available energy drink (16oz) + 2 pieces of placebo gum
  Interventions: Other: energy drink; Other: placebo gum
- Caffeinated drink and placebo gum (Active Comparator): Commercially-available caffeinated drink (16oz) + 2 pieces of placebo gum
  Interventions: Other: caffeinated drink; Other: placebo gum
- Control drink and energy gum (Active Comparator): Control drink (16oz) + 2 pieces of energy gum
  Interventions: Other: Energy gum; Other: Control drink
- Control drink and placebo gum (Placebo Comparator): Control drink (16oz) + 2 pieces of placebo gum
  Interventions: Other: placebo gum; Other: Control drink
- Energy drink and total sleep deprivation (Active Comparator): Commercially-available energy drink (16oz) + 2 pieces of placebo gum following total sleep deprivation
  Interventions: Other: energy drink; Other: placebo gum; Other: Total sleep deprivation

INTERVENTIONS:
Other: energy drink — 16 oz cold commercially-available energy drink
  Arms: Energy drink and placebo gum; Energy drink and total sleep deprivation
Other: caffeinated drink — 16oz cold commercially-available caffeinated drink
  Arms: Caffeinated drink and placebo gum
Other: Energy gum — 2 pieces of commercially-available energy gum
  Arms: Control drink and energy gum
Other: placebo gum — 2 pieces of commercially-available placebo gum
  Arms: Caffeinated drink and placebo gum; Control drink and placebo gum; Energy drink and placebo gum; Energy drink and total sleep deprivation
Other: Control drink — 16oz cold control drink
  Arms: Control drink and energy gum; Control drink and placebo gum
Other: Total sleep deprivation — 24-hour total sleep deprivation prior to consumption of energy drink and placebo gum
  Arms: Energy drink and total sleep deprivation

SUMMARY:
The purpose of this study will be to examine the acute effect of commercially available energy products on endothelial function, arterial stiffness and thrombosis in healthy young males.

DETAILED DESCRIPTION:
The use of energy products has significantly increased in the last few years and is especially high among young men. The present study will compare the acute effect of a commercially available energy drink, energy gum, coffee and control beverage on endothelial function, arterial stiffness and circulating markers of thrombosis, inflammation and oxidative stress.

ELIGIBILITY:
Inclusion Criteria:

* Being Male
* 18-30 years of age
* No indication of major clinical disease (e.g. diabetes, hypertension, significant arrhythmias, syncope and cardiovascular disease)
* BMI ≤ 30 kg/m^2 and blood pressure ≤ 140/90 mmHg
* Consumption of <400mg of caffeine/day
* Prior history of consumption of energy drinks

Exclusion criteria:

* Being female
* Age <18 or >30 years
* BMI> 30 kg/m^2 and blood pressure > 140/90 mmHg
* Use of medication that may affect vascular measures
* Use of tobacco products including smoking
* Vegan or vegetarian diet
* Being energy drink or caffeine naïve or consumption of >400 mg of caffeine/day
* Consumption of >1 energy drinks per month
* Being a shift worker

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2018-01-12 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-05-16 (Actual)

PRIMARY OUTCOMES:
Change in endothelial function | Before and 1 and 2 hrs following consumption of drink and gum
  Brachial artery flow-mediated dilation

SECONDARY OUTCOMES:
Change in arterial stiffness | Before and 1 and 2 hrs following consumption of drink and gum
  Carotid to femoral pulse wave velocity
Change in wave reflection | Before and 1 and 2 hrs following consumption of drink and gum
  Augmentation index
Change in peripheral and central blood pressures | Before and 1 and 2 hrs following consumption of drink and gum
  Brachial and aortic blood pressures
Change in thrombosis and platelet function | Before and 1 and 2 hrs following consumption of drink and gum
  Thromboelastograph and platelet aggregation tests
Change in circulating factors related to vascular function | Before and 1 and 2 hrs following consumption of drink and gum
  Circulating levels of Trimethylamine N-oxide (TMAO) and markers of oxidative stress and inflammation
Change in heart rhythm | Before and 1 and 2 hrs following consumption of drink and gum
  Electrocardiogram

CONTACTS AND LOCATIONS:
Overall Officials: Demetra Christou, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States